CLINICAL TRIAL: NCT05908110
Title: The Role of Health Communication Messaging in Evidence-based Pediatric Obstructive Sleep Apnea Detection
Brief Title: Evidence-based Pediatric Obstructive Sleep Apnea Detection
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Eskenazi Health (Other)
Responsible Party: Principal Investigator, Sarah Honaker, Associate Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 14456; K23HL150299-01 (NIH)
Record Dates: First submitted 2023-05-22; First posted 2023-06-18 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Obstructive Sleep Apnea of Child

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to: 1) intervention (seeing a health communication message about OSA) or 2) Usual care.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The primary care provider will receive the same alert for a positive OSA screen regardless of randomization condition. The primary outcome (OSA referral completion) will be extracted from the medical record by team members who are not aware of the child's randomization status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Communication Message (Experimental): Parents will review a health communication message (infographic) informing them that their child has OSA symptoms, describing both nighttime and daytime OSA symptoms, and encouraging them to speak to their child's primary care provider at the scheduled visit if they observe symptoms in their child. Primary care providers will receive an alert that the child screened positive for OSA.
  Interventions: Behavioral: Health Communication Message
- Usual Care (No Intervention): Like in the intervention group, parents will complete screening items and primary care providers will receive an alert if the child screens positive for OSA. However, parents randomized to this condition will not view the health communication message nor receive any information about OSA or their child's risk for OSA.

INTERVENTIONS:
Behavioral: Health Communication Message — The health communication message is a single infographic developed iteratively with input from stakeholders (parents and providers). This image informs the parent that their child may have OSA, lists common nighttime symptoms parents may observe (e.g., snoring, apnea) and common daytime symptoms (e.g., hyperactivity, sleepiness) that can result from OSA. Parents are then encouraged to speak to their child's primary care provider if they observe these symptoms in their child.
  Arms: Health Communication Message

SUMMARY:
The goal of this clinical trial is to test whether a health communication message (infographic about obstructive sleep apnea; OSA) seen by parents whose children have OSA symptoms will be helpful in identifying children with OSA. The main questions it aims to answer are:

* Will parents who see this health communication message be more likely to talk to their child's health care provider about OSA?
* Does the use of a health communication message help health care systems identify more children with OSA?

Participants are parents and children who are patients in a specific health care center. As part of clinical care, parents will answer screening questions about OSA symptoms (e.g., snoring, sleepiness) before their child's primary care visit. If their child has OSA symptoms, the health care provider will receive an alert suggesting further evaluation and possible referral for a sleep study or to a specialist.

In this study, children with OSA symptoms whose parents answer screening questions will be randomized to one of two conditions: 1) Health communication message (parent sees message before their child's visit with a primary care provider); or 2) Usual care (no information about OSA or their child's risk).

Researchers will compare groups to see if the health communication message helps identify more children with OSA.

DETAILED DESCRIPTION:
Many children with obstructive sleep apnea (OSA) are not identified and thus do not receive treatment. In a previous study, the investigators found that a clinical decision support system helped primary care providers (PCPs) identify children with obstructive sleep apnea (OSA). In this system, parents of children report on possible OSA symptoms (e.g., snoring, sleepiness) in their child before the visit. If the child has OSA symptoms, the PCP receives an alert during the visit recommending further evaluation and a possible referral for a sleep study or to see a specialist. While this system helped increase the number of children with OSA symptoms who received a referral, many children remained unidentified. The goal of this study is to see whether involving parents in the system can identify even more children.

In this study, the investigators propose to test the impact of a health communication message, designed to educate and activate parents about their child's risk for OSA. This message is an infographic that helps parents recognize nighttime symptoms of OSA and how these nighttime symptoms may be impacting their child during the day. If a child has OSA symptoms, parents would view this infographic before their child's PCP visit and could discuss OSA with their child's PCP. For children with OSA symptoms, their parents will be randomized to either: 1) view the health communication message, or; 2) usual care, in which parents are not given any additional information about OSA or their child's risk prior to the appointment. In both cases, PCPs will receive a prompt indicating that the child is at risk for OSA.

ELIGIBILITY:
Inclusion Criteria:

* Child ages 2.0-13.9 years at the time of OSA screening.
* Child is a primary care patient at Eskenazi Health
* Parent completed pre-visit questionnaire with OSA screening items
* Child screened positive for OSA (snoring >= 3 nights/wk + 1 additional symptom)

Exclusion Criteria:

* Prior OSA diagnosis
* Prior OSA referral (ENT, PSG, Sleep medicine) in the past two years

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2026-11-14 (Estimated); Study Completion 2026-11-14 (Estimated)

PRIMARY OUTCOMES:
Rate of Completed OSA referral | Up to 9 months after study entry (date of positive OSA screen)
  Rate of children who received and completed (e.g., attended appointment or sleep study) a referral for sleep-disordered breathing, amongst those who screened positive for OSA. Referrals to include: 1) polysomnogram; 2) ENT referral; or 3) sleep medicine referral.

SECONDARY OUTCOMES:
Rate of OSA referral | Up to 3 months after study entry (date of positive screen)
  Rate of children who received referral for sleep-disordered breathing, amongst whose who screened positive for OSA. Referrals to include: 1) polysomnogram; 2) ENT referral; or 3) sleep medicine referral.
Rate of Evidence-based Evaluation | Up to 3 months after study entry (date of positive screen)
  Rate of child who received evidence-based evaluation for pediatric OSA, amongst those who screened positive for OSA. Evidence-based evaluation includes 1) OSA referral; 2) documented watchful waiting with follow-up plan; and/or 3) documentation of evaluation not consistent with sleep-disordered breathing.
Rate of OSA Diagnosis | Up to 9 months after study entry (date of positive screen)
  Rate of children who received an OSA diagnosis (verified via polysomnogram; apnea hypopnea index >1.5), amongst those who screened positive for OSA.
Rate of OSA Treatment | Up to 12 months after study entry (date of positive screen)
  Rate of children receiving OSA treatment, amongst those who screened positive for OSA. Treatment to include 1) surgical intervention; 2) CPAP; 3) dental device; and/or 4) medication.
Rate of Parent Activation | Immediately after intervention (viewing the Health Communication Message)
  Rate of parents who report planning to speak with child's provider about OSA, amongst those who viewed the health communication message. This will be measured by parental response to an item asking if they plan to speak with their child's provider about OSA, presented at the time that the parent reviews the health communication message.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share data consistent with the requirements of the funder (NHLBI) and my institution.
Time Frame: Deidentified data will be available 1 year after study completion for a period of 5 years.
Access Criteria: By investigator request to the PI. Requesting investigator to submit description of research aims and analytic plan.